CLINICAL TRIAL: NCT05697822
Title: The Effect of a Patient-involved Mobile Phone and Cloud-based Electronic Contact and Recording System on Institutional Deliveries and Other Maternal and Infant Health Outcomes in Rural Nepal: A Cluster Randomized Controlled Trial
Brief Title: Using Advanced Data Systems to Improve Health in Early Life in Rural Nepal
Acronym: CITH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amit Arjyal (Other)
Collaborators: Bagmati Rural Municipality, Lalitpur, Nepal (Unknown); Konjyosom Rural Municipality, Lalitpur, Nepal (Unknown); Mahankal Rural Municipality, Lalitpur, Nepal (Unknown); School of Health Sciences, Purbanchal University, Nepal (Unknown)
Responsible Party: Sponsor-Investigator, Amit Arjyal, Assistant Professor, Patan Academy of Health Sciences
Organization: Patan Academy of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2-2022; CTSR - 77/78 - 4 (Other Grant/Funding Number: University Grants Commission - Nepal)
Record Dates: First submitted 2023-01-10; First posted 2023-01-26 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Maternal Health; Infant Health; Institutional Delivery; Birth Preparedness and Complication Readiness; Severe Maternal Morbidity; Neonatal Adverse Outcome
Keywords: electronic health database; maternal health; infant health; institutional delivery; birth preparedness and complication readiness; severe maternal morbidity; neonatal adverse outcome; mobile health; mHealth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is open-label as both the participants and study team members will know whether they are in the intervention or control arms. However, the outcomes related to morbidity will be assessed by a masked assessor.
  The outcomes such as severe maternal morbidity (SMM), and neonatal adverse outcomes(NAO) will be assessed by a study technical committee member who do not have any knowledge about the arm in which the study participant is allocated. The information about the study arm will be removed from the database when this assessment is being made. Although the criteria for SMM and NAO are generally objective, there might be some need for judgement on the part of the assessors hence masking will avoid biased assessment of outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Phone and Cloud-based Electronic Contact and Recording System (Experimental): In this arm pregnant women will be given a smart mobile-phone with an application installed which will have their detailed health-related information. They will be able to use this application to input their daily symptoms. This will also contain results of examinations or investigations that they have undergone in a clinic. All this information will be stored in a cloud and the healthcare worker at the local health post will also be able to access this information in their mobile phone and keep track of the pregnant women under their care. In the event of a concerning symptom, the health worker will be flagged. The health coordinators in the rural municipality will also be able to keep track of the pregnant women in their area through a cloud-based database.
  Interventions: Other: Mobile Phone and Cloud-based Electronic Contact and Recording System
- Usual Standard of Care Arm (No Intervention): Pregnant women will visit the health posts or hospitals for antenatal checks routinely as advised. Their records will be kept in paper-based forms and registers. They will not be tracked regularly by their healthcare provider by electronic means. Their daily symptoms will not be recorded anywhere. They will still be able to contact their healthcare providers or visit the health centers if necessary. They will not have a personal electronic health record. No one will keep active track of the pregnant women through electronic means.

INTERVENTIONS:
Other: Mobile Phone and Cloud-based Electronic Contact and Recording System — A mobile phone application has been developed which is intended to be used by pregnant women and their healthcare workers. A pregnant woman can get registered in this app and enter information and data related to their health and current pregnancy. Their health worker at their health post can access this information on their mobile phone too. The pregnant woman can also input her daily symptom on this app. She can also input and/or access information on examination and tests that have been carried out. If a concerning symptom or event has been entered by a user in the app, the health worker will be notified through this app. The health worker can also track the pregnant women under their care through this application. A cloud-based database of pregnant women will have the details of all the pregnant women in a given ward or rural municipality. Health coordinators in the municipality will be able to access the database for their municipality and track the pregnant women, if needed.
  Other Names: Mobile Phone Application
  Arms: Mobile Phone and Cloud-based Electronic Contact and Recording System

SUMMARY:
The goal of this cluster randomized controlled trial is to study the effect of a mobile-phone based application used by pregnant women on maternal and newborn health indicators. The main objective is to compare the rates of institutional deliveries in the intervention and control arms. Ancillary objectives are to compare the birth-preparedness and complication readiness parameters, severe maternal morbidity rates and neonatal adverse outcomes rates in the two arms. The participants are pregnant women.

In the intervention arm pregnant women will be given a smart mobile phone with an application that they will use to input information related to their health. This information can be shared with their healthcare workers. The healthcare workers will also be able to access all the health-related details of the pregnant women and mothers under their care by accessing this app in their mobile phones and be in touch with their patients through the mobile phone application.

The control arm will adhere to existing practices of pregnant woman and health worker communication without the use of a smart mobile phone with an existing application. Records related to the pregnant woman will be kept in paper-based forms as is the usual norm.

The investigators will compare the intervention arm and the control arm to see if there are differences in the rates of the outcomes.

DETAILED DESCRIPTION:
Improving maternal and newborn health requires innovative approaches that are flexible and cater to the need of the end-user, the patient. In the recent years telecommunication services that have seamlessly entered the lives of the both providers and receivers of health care both in developing and underdeveloped nations and have been a fertile ground for such innovations. There has been rapid growth of the use of mobile phone technologies (mobile health/mHealth) in low and middle income countries (LMICs). These function predominantly in the areas of client education and behavior change communication, registries and vital event tracking, data collection and reporting, provider to provider communication and electronic health records. In our setting as well, there has been successful implementation of the electronic medical records at health facility level and community based institutions and mobile health applications for the community level health providers. The major users of these digital platforms are service providers rather than patients.

However, using electronic medical records that a pregnant woman and/or a mother can fill up at home may provide more opportunities to identify risks and practices that reflect the real situation better than surveys or registries which rely on recall. So far, there is no such intervention in our setting to incorporate the users as the direct data keepers in the health system. Also, there is lack of evidence on the benefit of such applications for maternal and child health. Therefore, we are conducting a cluster randomized controlled trial on user based advanced data systems to improve health in early life in rural Nepal.

The intervention will be evaluated using a cluster randomized controlled trial design. The rationale is that the intervention is applied to the entire community and individual randomization is not feasible due to contamination. A rural municipality ward, the lowest administrative level in Nepal, will be randomized into intervention or control cluster. Because of the nature of the intervention, allocation is not masked. This project will be carried out in three rural municipalities of southern Lalitpur District, namely Konjyosom, Mahankal and Bagmati Rural Municipalities. Eighteen wards or clusters, nine(9) in the intervention arm and nine(9) in the control arm are included.

The investigators will implement the mobile-phone based system in the intervention clusters while non-intervention clusters will have the currently existing health care data management and patient contact system.

In the intervention arm, a data-system with mobile phone-based application will be deployed. The application will be used by pregnant women to obtain useful information related to their pregnancy and also enter vital information related to their health. The database will be accessible to healthcare providers at various levels of our health system such as health posts, and district or municipal level hospitals. The healthcare providers will also be able to access the data and enter clinical information when the pregnant women go to the health centre. The application will also be used during the time of labour and after delivery to record information about the post-partum state and infancy of the newborn child.

The investigators will carry out a prospective follow-up in which all institutional/home deliveries, birth preparedness and complication readiness parameters, severe maternal morbidity, neonatal adverse outcomes, stillbirths, neonatal and later infant deaths and deaths of women in the study population are recorded through interviews conducted during the recruitment, at 6-9 months of pregnancy, right after delivery and at 42 days after delivery.

This study is led by Patan Academy of Health Sciences, Lalitpur, Nepal in collaboration with Purbanchal University, Lalitpur, Nepal. The investigators have received a grant from University Grants Commission, Nepal for this project. The investigators have signed a Memorandum of Understanding with the three rural municipalities of southern Lalitpur namely, Bagmati, Konjyosom and Mahankal Rural Municipalities and plan to work in close liaison with the Ministry of Health, Department of Health Services, Health Office for Lalitpur District and Government Integrated Data centre (GIDC) to undertake this project.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with less than 20 weeks of gestation
* Usual resident of the study ward at the time of enrollment (A woman is considered a usual resident if the house she normally lives is in, is in that ward)
* Provides informed written consent

Exclusion Criteria:

* Temporary resident of the ward
* Cannot read and write
* Cannot use a mobile phone
* Has any disability, such as blindness, that prevents the use of mobile phone

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Institutional Delivery Rate | At the time of delivery
  Delivery at a birthing center, health post, primary health care center, or any hospital

SECONDARY OUTCOMES:
Birth Preparedness and Complication Readiness Index Score | Upto 42 days after delivery
  Birth preparedness and complication readiness index score will be used. It is based on JHPIEGO manual on monitoring birth preparedness and complication readiness- tools and indicators for maternal and newborn health. This is based on a set of indicators for monitoring safe motherhood. The final score is the average of thirteen(13) items in three(3) domains, namely, knowledge of key danger signs around pregnancy, service use and planning actions- both intention and behavior, and knowledge of community resources. A score will be calculated for each item as a percentage of the respondents who meet the item criteria. The final score is the mean of the scores in each of the 13 items. The score can range from 0% to 100%, higher score indicating better birth preparedness and complication readiness. The scores will be compared between the intervention and control arms.
Severe Maternal Morbidity (SMM) Rate | Upto 42 days after delivery
  Severe Maternal Morbidity criteria will be as defined by the American College of Obstetricians and Gynecologists (ACOG) criteria:
  1. The occurrence of at least one of 21 SMM indicators: Acute Myocardial Infarction, Aneurysm, Acute renal failure, Adult respiratory distress syndrome, Amniotic fluid embolism, Cardiac arrest/ ventricular fibrillation, Conversion of cardiac rhythm, Disseminated Intravascular coagulation, Eclampsia, Heart Failure/Arrest during surgery or procedure, Puerperal cerebrovascular disorders, Pulmonary edema/ Acute heart failure, Severe anesthesia complication, Sepsis, Shock, Sickle cell disease with crisis, Air and thrombotic embolism, Blood product transfusion, Hysterectomy, Temporary tracheostomy and Ventilation.
  2. Intensive care unit (ICU) admission
  3. Prolonged length of postnatal hospital stay (> 48 hours and >96 hours for vaginal delivery and cesarean section respectively)
  4. Transfusion of >/= 4 units of packed blood cells
  5. Hospital readmission
Neonatal Adverse Outcome (NAO) Rate | Upto 42 days after delivery
  NAO will be defined as the occurrence of at least one of 28 diagnostic and procedure components:
  Diagnosis: Gestational age < 32 weeks, birthweight <1500 grams, death within 28 days of birth, Birth trauma, Cerebral conditions like: Intraventricular haemorrhage, Hypoxic-ischemic encephalopathy, seizures, or other cerebral diagnosis, Respiratory conditions like: Pneumonia, Respiratory distress syndrome, Bronchopulmonary dysplasia and Other respiratory diagnosis, Sepsis/septicaemia, Necrotising enterocolitis Procedure: Resuscitation or intubation recorded on birth record, Transferred to higher center within 24 hours, 2-999 hours of mechanical ventilation, Invasive ventilation procedure, Non-invasive ventilation procedure, Resuscitation procedure, Arterial/central catheter procedure, Transfusion of blood or blood products, Intravenous fluid procedure, Surgical procedures: Abdominal, cardiac, thoracic and urinary system
Newborn Mortality Indicators | Upto 42 days after delivery
  Number of still births, early and late neonatal mortality, or infant mortality
Maternal Mortality Indicator | Upto 42 days after delivery
  Number of maternal deaths

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan P Devbhandari, MBBS,PhD, Principal Investigator — Patan Academy of Health Sciences
Locations (1):
- Patan Academy of Health Sciences, Lalitpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
When the dataset is available we will decide in what form we will share it with other researcher after determining their objective

REFERENCES:
- [Background] Del Barco R, editor. JHPIEGO Monitoring Birth Preparedness and Complication Readiness, Tools and Indicators for Maternal and Newborn Health. Baltimore (USA): JHPIEGO; 2004. Available from: https://pdf.usaid.gov/pdf_docs/Pnada619.pdf
- [Background] Main EK, Abreo A, McNulty J, Gilbert W, McNally C, Poeltler D, Lanner-Cusin K, Fenton D, Gipps T, Melsop K, Greene N, Gould JB, Kilpatrick S. Measuring severe maternal morbidity: validation of potential measures. Am J Obstet Gynecol. 2016 May;214(5):643.e1-643.e10. doi: 10.1016/j.ajog.2015.11.004. Epub 2015 Nov 12. PMID 26582168
- [Background] Callaghan WM, Creanga AA, Kuklina EV. Severe maternal morbidity among delivery and postpartum hospitalizations in the United States. Obstet Gynecol. 2012 Nov;120(5):1029-36. doi: 10.1097/aog.0b013e31826d60c5. PMID 23090519
- [Background] Nam JY. Comparison of global indicators for severe maternal morbidity among South Korean women who delivered from 2003 to 2018: a population-based retrospective cohort study. Reprod Health. 2022 Aug 13;19(1):177. doi: 10.1186/s12978-022-01482-y. PMID 35964088
- [Background] Todd S, Bowen J, Ibiebele I, Patterson J, Torvaldsen S, Ford F, Nippita M, Morris J, Randall D. A composite neonatal adverse outcome indicator using population-based data: an update. Int J Popul Data Sci. 2020 Aug 12;5(1):1337. doi: 10.23889/ijpds.v5i1.1337. PMID 33644407
- [Background] Huda TM, Chowdhury M, El Arifeen S, Dibley MJ. Individual and community level factors associated with health facility delivery: A cross sectional multilevel analysis in Bangladesh. PLoS One. 2019 Feb 13;14(2):e0211113. doi: 10.1371/journal.pone.0211113. eCollection 2019. PMID 30759099
- [Background] Neupane B, Rijal S, Gc S, Basnet TB. A Multilevel Analysis to Determine the Factors Associated with Institutional Delivery in Nepal: Further Analysis of Nepal Demographic and Health Survey 2016. Health Serv Insights. 2021 Jun 14;14:11786329211024810. doi: 10.1177/11786329211024810. eCollection 2021. PMID 34177270
- [Background] Hemming K, Girling AJ, Sitch AJ, Marsh J, Lilford RJ. Sample size calculations for cluster randomised controlled trials with a fixed number of clusters. BMC Med Res Methodol. 2011 Jun 30;11:102. doi: 10.1186/1471-2288-11-102. PMID 21718530